CLINICAL TRIAL: NCT02971761
Title: A Phase 2 Clinical Trial of the Combination of Pembrolizumab and Selective Androgen Receptor Modulator (SARM) GTX-024 in Patients With Metastatic Androgen Receptor (AR) Positive Triple Negative Breast Cancer (TNBC)
Brief Title: Pembrolizumab and Enobosarm in Treating Patients With Androgen Receptor Positive Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16131; NCI-2016-01759 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16131 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2022-06-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Androgen Receptor Positive; Estrogen Receptor Negative; HER2/Neu Negative; Metastatic Triple-Negative Breast Carcinoma; Progesterone Receptor Negative; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — ostarine; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, enobosarm) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and enobosarm PO QD on days 1-21. Courses repeat every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enobosarm; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Enobosarm — Given PO
  Other Names: Gtx-024; Ostarine
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies the side effects and how well pembrolizumab and enobosarm work in treating patients with androgen receptor positive triple negative breast cancer that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Androgen can cause the growth of breast cancer cells. Hormone therapy using enobosarm may fight breast cancer by blocking the use of androgen by the tumor cells. Giving pembrolizumab and enobosarm may work better than pembrolizumab alone in treating patients with androgen receptor positive triple negative breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety/tolerability of the combination regimen. II. To determine the response rate (complete response [CR] or partial response [PR] via Response Evaluation Criteria in Solid Tumors [RECIST] 1.1) of the combination of pembrolizumab with enobosarm (GTx-024) in patients with advanced androgen receptor (AR) positive (+) triple negative breast cancer (TNBC).

SECONDARY OBJECTIVES:

I. To evaluate clinical outcomes by RECIST 1.1 including clinical benefit rate (CBR) at 24 weeks, progression free-survival (PFS), duration of response (DOR), event free survival (EFS), time-to-treatment failure (TTF); and overall survival (OS).

II. To evaluate the role of immune-related response criteria (irRECIST). III. To evaluate the association of AR by immunohistochemistry (IHC) and clinical response.

EXPLORATORY OBJECTIVES:

I. To evaluate the association of an AR gene expression signature and clinical response.

II. To evaluate genomic and phenotypic status of breast tumor. III. To evaluate the effect of the combination therapy on peripheral blood circulating tumor cells (CTCs) and circulating tumor deoxyribonucleic acid (DNA) (ctDNA).

IV. To evaluate the effect of combination therapy on tumor-derived exosomes (TEX) and TEX associated immune biomarkers.

V. Immune correlatives:

Va. To evaluate pre-treatment programmed death ligand 1 (PD-L1) and tumor infiltrating lymphocytes (TILs) as a predictor of response to combination therapy.

Vb. To evaluate specific TIL subsets (e.g. CD4, CD8, regulatory T cell [Treg] distribution) and other immunological correlatives (e.g. T cell receptor [TCR] repertoire analysis) as possible predictors of response.

Vc. To evaluate change in TILs as a result of the combination therapy. Vd. To evaluate peripheral blood, immune biomarkers.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and enobosarm orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days, every 3 months, and bi-annually.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent
* Willing to provide a sample from a recently obtained (within 42 days prior to initiation of day 1) biopsy of a tumor lesion

  * If recently-obtained samples are unavailable an archived metastatic specimen not previously irradiated may be submitted upon agreement from the study principal investigator (PI)
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Life expectancy of > 3 months
* Metastatic triple negative breast cancer (TNBC)
* Measurable disease per RECIST version (v)1.1 criteria: at least 1 lesion of > 10 mm in long axis diameter for non-lymph nodes or > 15 mm in short axis diameter for lymph nodes that is serially measurable according to RECIST 1.1 using computerized tomography, magnetic resonance imaging, or panoramic and close-up color photography
* Histologically proven diagnosis of TNBC per current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guideline

  * Estrogen receptor (ER) negative (ER expression =< 10% positive tumor nuclei), progesterone receptor (PR) negative (PR expression =< 10% positive tumor nuclei) and HER2 negative breast cancer by IHC and /or fluorescence in situ hybridization (FISH)
* Androgen receptor positive (AR+)

  * Defined as >= 50% nuclear AR staining by immunohistochemistry (IHC) in either the primary or metastatic lesion
  * NOTE: research testing of AR status is available at City of Hope (COH) Pathology
* Resolution of grade 2 and above toxicities of most recent therapy except for stable sensory neuropathy (=< grade 2) and alopecia
* Female (childbearing potential): use an adequate method of birth control (except hormonal contraception) or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication

  * Childbearing potential defined as not being surgically sterilized or have not been free from menses for > 1 year
* Male: use and adequate method of contraception with the first dose of study therapy through 120 days after the last dose of study therapy

  * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Absolute neutrophil count (ANC) >= 1500/mm^3 (within 14 days prior to day 1 of protocol therapy)
* Platelets >= 100,000/mm^3 (within 14 days prior to day 1 of protocol therapy)
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment) (within 14 days prior to day 1 of protocol therapy)
* Serum total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN if total bilirubin levels > 1.5 x ULN (within 14 days prior to day 1 of protocol therapy)
* Albumin >= 2.5 mg/dL (within 14 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN OR =< 5.0 x ULN if liver metastases present (within 14 days prior to day 1 of protocol therapy)
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (if measured or calculated per institutional standard; glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min if creatinine levels > 1.5 x ULN (within 14 days prior to day 1 of protocol therapy)
* Female of childbearing potential only: negative urine or serum pregnancy test; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required (within 14 days prior to day 1 of protocol therapy)

Exclusion Criteria:

* Anti-programmed cell death protein-1 (anti-PD-1), PD ligand-1 (PD-L1), PD ligand-2 (PD-L2) agent, an antibody targeting other immuno-regulatory receptors or mechanisms
* Radiotherapy within 14 days prior to day 1 of protocol therapy
* AR targeted agents (including GTx-024, enzalutamide or other AR targeted therapies)
* Investigational agent within 21 days prior to day 1 of protocol therapy
* Hormone replacement therapies (estrogens, megestrol acetate) within 14 days prior to day 1 of protocol therapy
* Live-virus vaccination within 30 days prior to day 1 of protocol therapy
* Systemic cytotoxic chemotherapy, antineoplastic biologic therapy, or major surgery within 21 days of the first dose of trial medication
* Testosterone or testosterone-like agents (methyltestosterone, oxandrolone, oxymetholone, danazol, fluoxymesterone, dehydroepiandrosterone, androstenedione) other androgenic compounds or anti-androgens within 30 days prior to day 1 of protocol therapy
* Chronic systemic steroid therapy or on any other form of immunosuppressive medication
* Unstable or untreated brain/leptomeningeal metastasis
* Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, or abdominal carcinomatosis (known risks factors for bowel perforation)
* Active central nervous system metastases and/or carcinomatous meningitis
* Severe hypersensitivity reaction to treatment with another monoclonal antibody
* Active autoimmune disease that has required systemic treatment in the past 2 years (replacement therapies for hormone deficiencies are allowed)
* Known history of human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* History of pneumonitis (non-infectious) that required steroids or current pneumonitis
* Diagnosed with or treated for cancer within the previous two years, other than breast cancer or non-melanoma carcinoma of the skin
* Unable to swallow capsules
* Currently on bisphosphonate or denosumab with elevated serum calcium levels corrected for albumin/ionized calcium levels outside of institutional normal limits
* Female: pregnant or lactating
* Concomitant medical condition that precludes adequate study treatment compliance or assessment, or increases subject risk, in the opinion of the investigator, such as but not limited to:

  * Myocardial infarction or arterial thromboembolic events within 6 months prior to baseline or severe or unstable angina, New York Heart Association (NYHA) class III or IV disease, or a QTCB (corrected according to Bazett's formula) interval > 470 msec; serious uncontrolled cardiac arrhythmia grade II or higher according to NYHA; uncontrolled hypertension (systolic > 150 and/or diastolic > 100 mm Hg)
  * Acute and chronic active infectious disorders and non-malignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this study therapy
  * Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2022-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Yuan, Principal Investigator — City of Hope Medical Center
Locations (7):
- United States (7):
  - City of Hope Corona, Corona, California
  - City of Hope Medical Center, Duarte, California
  - City of Hope Antelope Valley, Lancaster, California
  - City of Hope Mission Hills, Mission Hills, California
  - City of Hope Rancho Cucamonga, Rancho Cucamonga, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope West Covina, West Covina, California

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients seen at the City of Hope main campus and its surrounding affiliated community clinics.
Pre-assignment Details: Study was conducted from June 1, 2017 to October 28, 2019.
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
Started | 18
Completed | 16
Not Completed | 2
Not completed — GTx-024 drug supply was withdrawn | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 64 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic White | 8
  Hispanic | 5
  Asian | 2
  African American | 1
Region of Enrollment [Number; unit: participants]
  United States | 16
Number of previous lines of therapy [Count of Participants; unit: Participants]
  Received 0-1 previous lines of therapy | 9
  Received >=2 previous lines of therapy | 7
Performance Status (ECOG) [Count of Participants; unit: Participants] — Stage 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    ECOG stage 0 | 7
    ECOG stage 1 | 9
Nottingham Histological grade [Count of Participants; unit: Participants] — Nottingham Histologic Grade (Elston-Ellis modification of Scharff-Bloom-Richardson grading system). Higher grades have tissue histologies that are more involved with cancer.
  Participants
    Grade 1 | 2
    Grade 2 | 5
    Grade 3 | 9
Initial tumor stage [Count of Participants; unit: Participants] — Stages are per American Joint Committee on Cancer (AJCC) staging version 7.0. Stage III is a more advanced diagnosis than Stage II, which is in turn more advanced than Stage I.
  Participants
    Stage I | 6
    Stage II | 8
    Stage III | 2
Prior surgery [Count of Participants; unit: Participants]
  Lumpectomy | 7
  Mastectomy | 9
Prior radiation [Count of Participants; unit: Participants]
  Yes, received prior radiation | 15
  No | 1

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete Response or Partial Response)
Description: Response rate (complete response or partial response) assessed using Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: Up to 36 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
Number analyzed (Participants) | 16
Participants
  Complete response | 1
  Partial response | 1
  Stable disease | 2
  Progressive disease | 12

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival assessed using Response Evaluation Criteria in Solid Tumors version 1.1. Kaplan-Meier estimates will be generated.
Time Frame: Time to disease progression/relapse or death as a result of any cause, assessed up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
Number analyzed (Participants) | 16
months | 2.6 [1.9 to 3.1]

3. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate assessed by immune-related Response Evaluation Criteria in Solid Tumors version 1.1.
Time Frame: At 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
Number analyzed (Participants) | 16
Participants | 4

4. Secondary Outcome: Overall Survival
Description: Overall survival assessed by Response Evaluation Criteria in Solid Tumors version 1.1. Kaplan-Meier estimates will be generated.
Time Frame: Time to death as a result of any cause, assessed up to 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
Number analyzed (Participants) | 16
months | 25.5 [10.4 to 30.9]

5. Secondary Outcome: Progression-free Survival
Description: Progression-free survival defined as failure of treatment or death as a result of any cause assessed by Response Evaluation Criteria in Solid Tumors version 1.1. Kaplan-Meier estimates will be generated.
Time Frame: Up to 1 year
Population: Two patients were not evaluable for response, and were excluded from progression-free survival.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
Number analyzed (Participants) | 16
months | 2.6 [1.9 to 3.1]

ADVERSE EVENTS:
Time Frame: 36 months from commencement of treatment
Arm/Group | Treatment (Pembrolizumab, Enobosarm)
All-Cause Mortality (participants affected / at risk) | 8/18
Serious Adverse Events (participants affected / at risk) | 4/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Enobosarm) (N=18)
10019279-Heart failure (Cardiac disorders) | 1 (1)
10021038-Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
10016750-Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
10001409-Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, Enobosarm) (N=18)
10002272-Anemia (Blood and lymphatic system disorders) | 5 (5)
10033557-Palpitations (Cardiac disorders) | 1 (1)
10040741-Sinus bradycardia (Cardiac disorders) | 1 (1)
10040752-Sinus tachycardia (Cardiac disorders) | 5 (5)
bradypnea (Cardiac disorders) | 1 (1)
10014020-Ear pain (Ear and labyrinth disorders) | 1 (1)
10001367-Adrenal insufficiency (Endocrine disorders) | 1 (1)
10020850-Hyperthyroidism (Endocrine disorders) | 1 (1)
10021114-Hypothyroidism (Endocrine disorders) | 1 (1)
10005886-Blurred vision (Eye disorders) | 1 (1)
eye discomfort (Eye disorders) | 1 (1)
10000060-Abdominal distension (Gastrointestinal disorders) | 1 (1)
10000081-Abdominal pain (Gastrointestinal disorders) | 3 (3)
10005265-Bloating (Gastrointestinal disorders) | 3 (3)
10010774-Constipation (Gastrointestinal disorders) | 5 (5)
10012318-Dental caries (Gastrointestinal disorders) | 1 (1)
10012727-Diarrhea (Gastrointestinal disorders) | 8 (8)
10013781-Dry mouth (Gastrointestinal disorders) | 1 (1)
10013946-Dyspepsia (Gastrointestinal disorders) | 1 (1)
10013950-Dysphagia (Gastrointestinal disorders) | 2 (2)
10015388-Esophageal pain (Gastrointestinal disorders) | 1 (1)
10016766-Flatulence (Gastrointestinal disorders) | 2 (2)
10017999-Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
10028813-Nausea (Gastrointestinal disorders) | 6 (6)
10047700-Vomiting (Gastrointestinal disorders) | 6 (6)
discomfort (Gastrointestinal disorders) | 1 (1)
10008531-Chills (General disorders) | 2 (2)
10011914-Death NOS (General disorders) | 4 (4)
10014222-Edema face (General disorders) | 1 (1)
10016059-Facial pain (General disorders) | 2 (2)
10016256-Fatigue (General disorders) | 13 (13)
10016558-Fever (General disorders) | 2 (2)
10017577-Gait disturbance (General disorders) | 1 (1)
10022095-Injection site reaction (General disorders) | 1 (1)
10033371-Pain (General disorders) | 3 (3)
10050068-Edema limbs (General disorders) | 4 (4)
10062466-Localized edema (General disorders) | 3 (3)
10062501-Non-cardiac chest pain (General disorders) | 4 (4)
DROWSINESS (General disorders) | 1 (1)
10001718-Allergic reaction (Immune system disorders) | 1 (1)
10005047-Bladder infection (Infections and infestations) | 1 (1)
10046300-Upper respiratory infection (Infections and infestations) | 3 (3)
10046571-Urinary tract infection (Infections and infestations) | 3 (3)
10048038-Wound infection (Infections and infestations) | 1 (1)
stomach flu (Infections and infestations) | 1 (1)
10016173-Fall (Injury, poisoning and procedural complications) | 2 (2)
10041569-Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
10001551-Alanine aminotransferase increased (Investigations) | 4 (4)
10003481-Aspartate aminotransferase increased (Investigations) | 4 (4)
10008661-Cholesterol high (Investigations) | 2 (2)
10011368-Creatinine increased (Investigations) | 1 (1)
10025256-Lymphocyte count decreased (Investigations) | 1 (1)
10029366-Neutrophil count decreased (Investigations) | 1 (1)
10035528-Platelet count decreased (Investigations) | 2 (2)
10047896-Weight gain (Investigations) | 2 (2)
10047900-Weight loss (Investigations) | 2 (2)
10049182-White blood cell decreased (Investigations) | 1 (1)
10002646-Anorexia (Metabolism and nutrition disorders) | 4 (4)
10020639-Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
10020647-Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
10020943-Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
10020949-Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
10021005-Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
10021018-Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
10021028-Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
10021038-Hyponatremia (Metabolism and nutrition disorders) | 5 (5)
10021059-Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
INCREASED TRIGLYCERIDES (Metabolism and nutrition disorders) | 1 (1)
10003239-Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
10003988-Back pain (Musculoskeletal and connective tissue disorders) | 6 (6)
10006002-Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
10008496-Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
10016750-Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
10028411-Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
10028836-Neck pain (Musculoskeletal and connective tissue disorders) | 4 (4)
10033425-Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
10062572-Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
GENERALIZED MSK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
LEFT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
RIGHT HIP PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
RIGHT KNEE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
RIGHT THIGH PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
increased muscle mass (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1)
muscle spasms (back) (Musculoskeletal and connective tissue disorders) | 1 (1)
actinic keratosis, hyperplastic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6)
10013573-Dizziness (Nervous system disorders) | 4 (4)
10013911-Dysgeusia (Nervous system disorders) | 1 (1)
10019211-Headache (Nervous system disorders) | 9 (9)
10020765-Hypersomnia (Nervous system disorders) | 1 (1)
10024264-Lethargy (Nervous system disorders) | 1 (1)
10034620-Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
10041349-Somnolence (Nervous system disorders) | 1 (1)
10044565-Tremor (Nervous system disorders) | 2 (2)
10002855-Anxiety (Psychiatric disorders) | 4 (4)
10012378-Depression (Psychiatric disorders) | 2 (2)
10022437-Insomnia (Psychiatric disorders) | 5 (5)
10024419-Libido decreased (Psychiatric disorders) | 1 (1)
10019450-Hematuria (Renal and urinary disorders) | 2 (2)
10037032-Proteinuria (Renal and urinary disorders) | 4 (4)
10046539-Urinary frequency (Renal and urinary disorders) | 1 (1)
10046593-Urinary urgency (Renal and urinary disorders) | 1 (1)
10061574-Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
10063057-Cystitis noninfective (Renal and urinary disorders) | 1 (1)
oliguria (mild) (Renal and urinary disorders) | 1 (1)
10006298-Breast pain (Reproductive system and breast disorders) | 1 (1)
10046904-Vaginal dryness (Reproductive system and breast disorders) | 1 (1)
10003504-Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10011224-Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
10013963-Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
10015090-Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10021143-Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
10028735-Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10035598-Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
10036402-Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10036790-Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
10041367-Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
10047924-Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
OBSTRUCTIVE PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
rhonchi breath sounds (Respiratory, thoracic and mediastinal disorders) | 1 (1)
10001760-Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
10013786-Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
10020642-Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
10033474-Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
10037087-Pruritus (Skin and subcutaneous tissue disorders) | 4 (4)
10037847-Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (3)
10037868-Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
10054541-Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
stent placement (Surgical and medical procedures) | 1 (1)
10016825-Flushing (Vascular disorders) | 1 (1)
10020407-Hot flashes (Vascular disorders) | 2 (2)
10020772-Hypertension (Vascular disorders) | 12 (12)
10021097-Hypotension (Vascular disorders) | 5 (5)
10025233-Lymphedema (Vascular disorders) | 2 (2)
10042554-Superficial thrombophlebitis (Vascular disorders) | 1 (1)
10043565-Thromboembolic event (Vascular disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
The trial was stopped early because of the withdrawal of GTx-024 drug supply. Full assessment of activity could not be completed as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/61/NCT02971761/Prot_SAP_000.pdf